CLINICAL TRIAL: NCT01402778
Title: Fixation of Thoracic Epidural Catheters Influencing Catheter-related Infections and Dislocation
Brief Title: Fixation of Thoracic Epidurals Influencing Catheter-related Infections and Dislocation
Acronym: TDPAFD
Status: Completed | Type: Observational
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Collaborators: University of Osnabrueck (Other)
Responsible Party: Principal Investigator, Klinik für Anästhesiologie, Prof. Dr. Peter Kienbaum, Heinrich-Heine University, Duesseldorf
Other Study IDs: 02-VBTSPK-2011
Record Dates: First submitted 2011-01-12; First posted 2011-07-26 (Estimated); Last update posted 2011-12-20 (Estimated); Status verified 2011-12

CONDITIONS: Dislocation; Infection; Line Colonisation; Line Insertion Site
MeSH Terms: conditions — Joint Dislocations; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cather fixation by tunneling and suture
- Catheter fixation by adhesive tape

SUMMARY:
Major interest in our investigation is to find out whether distinct fixation techniques influence catheter dislocation and/ or incidence of local inflammation. A systematic comparison of two different fixation techniques with regard to catheter location, analgetic potential and signs of local inflammation will be conducted. To ensure identical patients groups allocation will be strictly randomized. Furthermore, both patient groups will receive identical pain medication via the peridural catheter in situ. All catheter tips will be screened microbiologically after removal.

ELIGIBILITY:
Inclusion Criteria:

Patients aged > 18 years and operation with thoracic epidural

Exclusion Criteria:

Refusal of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged > 18 years
Sampling Method: Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2011-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Changes in catheter position | 4-6 days
  Difference in catheter position between day of insertion and day of removal, measured in mm between catheter tip and skin niveau

SECONDARY OUTCOMES:
Secondary variables | 4-6 days
  Analgetic quality, incidence of catheter contamination, signs of local inflammmation and microbiological eamination of the catheter after removal

CONTACTS AND LOCATIONS:
Overall Officials: Peter Kienbaum, Professor, Principal Investigator — Heinrich Heine University, Department of Anaesthesiology, Chairman: Univ-Prof. Dr.med. B. Pannen; Martin Beiderlinden, Privatdozent, Principal Investigator — Department of Anaesthesia, Marienhospital Osnabrueck
Locations (1):
- Heinrich Heine University, University Hospital Duesseldorf, Department of Anaesthesiology, Düsseldorf, North Rhine-Westphalia, Germany